CLINICAL TRIAL: NCT01148277
Title: Propofol and Remifentanyl Versus Midazolam and Fentanyl for Diagnostic Colonoscopy in Patients With Compensated Cirrhosis Child A-B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Liver Clinic, Ziv medical center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Propofol vs Midazolam
Record Dates: First submitted 2010-06-13; First posted 2010-06-22 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2010-06

CONDITIONS: Liver Disease
Keywords: Endoscopies; Liver diseases; Propofol; Midazolam and remifentanyl
MeSH Terms: conditions — Liver Diseases | interventions — Propofol; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Propofol and Remifentanyl (Active Comparator): Propofol, colonoscopies, liver diseases, cirrhosis
  Interventions: Drug: Propofol and Remifentnyl
- midazolam and fentanyl (Active Comparator): midazolam and fentanyl, colonoscopies, liver diseases
  Interventions: Drug: midazolam and fentanyl
- control midazolam anf fentanyl (Experimental): midazolam anf fentanyl
  Interventions: Drug: midazolam anf fentanyl

INTERVENTIONS:
Drug: Propofol and Remifentnyl — Intervention group (Propofol and remifentanyl): It will be administered under direct gastroenterologists' and hepatologist
  Arms: Propofol and Remifentanyl
Drug: midazolam and fentanyl — Intervention group (Propofol and fentanyl ): It will be administered under direct gastroenterologists'and hepatologist
  Arms: midazolam and fentanyl
Drug: midazolam anf fentanyl — group (Midazolam with Fentanyl): Both drugs will be administered by the gastroenterologists and/ or hepatologist and/ or anesthiologist
  Arms: control midazolam anf fentanyl

SUMMARY:
This is a prospective, randomized-controlled trial (RCT) comparing the use of Propofol and Remifentanyl and traditional sedation (Midazolam and Fentanyl) for diagnostic colonoscopies in patients with compensated cirrhosis child A-B. The working hypothesis is that the use of propofol will be translated in a shorter recovery and discharge times with a higher patient satisfaction and a decrease in general complications (Hepatic Encephalopathy) in the context of patients with advanced liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients older than 18 and younger than 75 years with cirrhosis defined by the presence of liver fibrosis at least F3 and higher in the METAVIR score or with established cirrhosis (Child Pugh A, B)

Exclusion Criteria:

* Patients with significant cardiorespiratory disease i.e. advanced respiratory, renal and heart failure (ASA class III or higher except for patients with decompensate liver cirrhosis), obstructive sleep apnea.
* HCC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of propofol in liver diseases | up to 3 hours
  At the end of each endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv medical center liver unit, Safed, Israel, Israel